CLINICAL TRIAL: NCT03389061
Title: Bioequivalence Study of Crushed Sofosbuvir/Velpatasvir Compared to the Whole Tablet
Acronym: CRUSADE-1
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of patients who are eligible for inclusion: less patients on treatment and not using epclusa.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF 16.06
Record Dates: First submitted 2017-09-25; First posted 2018-01-03 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: HCV
Keywords: Epclusa; Pharmacokinetics; Crushing
MeSH Terms: conditions — Pressure Ulcer | interventions — sofosbuvir-velpatasvir drug combination; Sofosbuvir

STUDY DESIGN:
Intervention Model Description: Bio-equivalence Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sofosbuvir/velpatasvir tablet (Active Comparator): Single-dose sofosbuvir/velpatasvir as a whole tablet in a fasted state.
  Interventions: Drug: sofosbuvir/velpatasvir tablet
- sofosbuvir/velpatasvir crushed (Experimental): Single-dose crushed sofosbuvir/velpatasvir in a fasted state.
  Interventions: Drug: sofosbuvir/velpatasvir crushed

INTERVENTIONS:
Drug: sofosbuvir/velpatasvir tablet — Single-dose SOF/VEL as a whole tablet in a fasted state.
  Arms: sofosbuvir/velpatasvir tablet
Drug: sofosbuvir/velpatasvir crushed — Single-dose crushed SOF/VEL in a fasted state.
  Arms: sofosbuvir/velpatasvir crushed

SUMMARY:
Epclusa® is a pan-genotypic, once-daily tablet for the treatment of chronic hepatitis C virus (HCV) infection containing the NS5B- polymerase inhibitor sofosbuvir (SOF, nucleotide analogue) 400 mg and the NS5A inhibitor velpatasvir (VEL) 100 mg.

For patients with swallowing difficulties, administration of whole tablets can be problematic. In addition, HCV patients that are hospitalized (at intensive care units) due to severe illness (co-infections/ liver failure) might not be able to swallow medication. Therefore it is useful to know whether it is possible to administer SOF/VEL through a different route, like a feeding tube.

In daily practice, information about the safety and efficacy of crushed tablets is lacking which might result in interruption or discontinuation of expensive HCV therapy. However, it is not recommended to interrupt treatment because there is no evidence about the efficacy of the therapy after discontinuation (and restart).

Currently, patients and healthcare professionals are crushing SOF/VEL tablets without information about efficacy and safety. Depending on the biopharmaceutical characteristics of a drug formulation, crushing tablets can lead to altered pharmacokinetics of drugs.

It is important to know whether pharmacokinetic parameters are influenced by crushing of tablets; both a decrease and an increase in exposure may occur. A decrease of the plasma concentrations of SOF and/or VEL potentially reduces the therapeutic effect of the drugs. Higher doses or switching to other HCV-drugs might be needed. In contrast, in case a higher Cmax,ss and/or exposure occurs there might be an increased risk of toxicity.

As a result, crushing the drug is a contra-indication based on the available data.

Therefore this study will be conducted to investigate whether a crushed SOF/VEL tablet is bioequivalent to SOF/VEL as a whole tablet.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with SOF/VEL treatment for the treatment of chronic HCV genotype 1 through 6.
2. Patient is at least 18 at the day of screening.
3. Patient is able and willing to sign the Informed Consent Form.
4. Patient is able and willing to follow protocol requirements.

Exclusion Criteria:

1. Pregnant female (as confirmed by an hCG urine test performed at screening) or breast-feeding female.
2. Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
3. Inability to understand the nature and extent of the study and the procedures required.
4. Clinically relevant low hemoglobin concentration at screening judged by the patient's own hepatologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
AUC | Up to 24 hours after administration
Cmax | one dosing interval after administration of SOF/VEL (up to 24 hours)

SECONDARY OUTCOMES:
Adverse events | During the entire conduct of the study, maximum of two weeks

CONTACTS AND LOCATIONS:
Locations (3):
- University of Bonn, Germany, Bonn, Germany
- Netherlands (2):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Radboud university medical center Department of GI tract, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Seyen M, Samson AD, Cullen L, Eastick K, Knol H, Colbers A, Burger DM. Crushed application of sofosbuvir and velpatasvir in a patient with swallowing disorder. Int J Antimicrob Agents. 2020 Jun;55(6):105934. doi: 10.1016/j.ijantimicag.2020.105934. Epub 2020 Mar 7. No abstract available. PMID 32156618